CLINICAL TRIAL: NCT02686827
Title: A Randomized, Double-blind, Placebo-controlled Study to Determine the Immune Effects of Multiple Doses of Vitamin D3 in Patients With Allergic Rhinitis/Rhino-conjunctivitis Caused by Birch Pollen and in Healthy Control Subjects.
Brief Title: DBPC-Dose-finding-trial of Vitamin D3 for SCIT in Birch Pollen Allergic Patients.
Acronym: BM4SIT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Laurian Jongejan (Other)
Responsible Party: Sponsor-Investigator, Laurian Jongejan, Project manager, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Organization: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: BM4SIT
Record Dates: First submitted 2016-01-28; First posted 2016-02-22 (Estimated); Last update posted 2018-09-04 (Actual); Status verified 2018-08

CONDITIONS: Hypersensitivity
MeSH Terms: conditions — Hypersensitivity | interventions — paricalcitol; Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Paricalcitol (Vitamin D3) (Experimental): paricalcitol, (Zemplar® 5 μg/ml Abbvie), will be administered via the subcutaneous route 4 times at 0.5 ml (registered dose of 5 μg/ml, thus 2.5 μg per sub-cutaneous injection). The minimum time interval between two injections is 4 days, which is a significantly lower frequency than the prescribed maximum of 3 times a week or every other day.
  Interventions: Drug: Paricalcitol
- Placebo (Active Comparator): Placebo, the same constituents as Zemplar (propylene glycol 30% (v/v) alcohol 20% (v/v)) but no paricalcitol, same dosage as verum-arm.
  Interventions: Drug: Placebo (for paricalcitol)

INTERVENTIONS:
Drug: Paricalcitol — Vitamin D3 analogue
  Other Names: Vitamin D3, (Zemplar)
  Arms: Paricalcitol (Vitamin D3)
Drug: Placebo (for paricalcitol) — Injection fluid to mimic paricalcitol injection
  Other Names: fluid to mimic paricalcitol injection
  Arms: Placebo

SUMMARY:
Low Vitamin D3 (VD3) levels have been reported to be associated with the risk of allergic diseases like asthma. VD3 has been demonstrated in vitro, ex vivo and in animal models to program the immune system towards anti-inflammatory immune responses. VD3 co-administered with allergen may be a promising adjuvant to improve the onset and efficacy of allergen immunotherapy (AIT). A clinical trial will be performed to compare the immune effects, the tolerability and safety of multiple doses of aVD3 analogue (registered for the intravenous route) administered by the subcutaneous (s.c.) route in subjects with allergic rhinitis and healthy controls.

The overall aim is to provide additional (in vivo) support for the use of VD3 as an adjuvant in allergen-specific immunotherapy, on top of the existing pre-clinical evidence demonstrating that antigen-presenting cells educate the adaptive immune system towards an anti-inflammatory response when allergen is seen in the presence of VD3.

DETAILED DESCRIPTION:
Low Vitamin D3 (VD3) levels have been reported to be associated with the risk of allergic diseases like asthma. In addition, VD3 has been demonstrated in vitro, ex vivo (skin-explants) and in animal models to program the immune system towards anti-inflammatory immune responses, dominated by regulatory T-cells (Treg) producing Interleukin (IL)-10. In response to allergens, healthy individuals by default have such a protective immune response against innocuous allergens, whereas allergic subjects develop an inflammatory Th2-type response. VD3 co-administered with allergen may be a promising adjuvant to improve the onset and efficacy of allergen immunotherapy (AIT), by helping the allergic immune system to divert towards an allergen-specific response dominated by regulatory T cells (Treg) and IL-10. A clinical trial will be performed to compare the immune effects, the tolerability and safety of multiple doses of a VD3 analogue (Zemplar® 5 μg/ml - Abbvie, registered for the intravenous route) administered by the subcutaneous (s.c.) route in subjects with allergic rhinitis and healthy controls. Primary and secondary outcomes will be compared at baseline and at several time points during the study to investigate whether 1) the healthy controls at baseline have a more anti-inflammatory systemic cellular immune response to polyclonal stimuli and to allergens compared to birch pollen allergic subjects, and 2) whether s.c.VD3 analogue can skew these responses in allergic subjects towards a profile more resembling the one observed in healthy controls. The overall aim is to provide additional (in vivo) support for the use of VD3 as an adjuvant in allergen-specific immunotherapy, on top of the existing pre-clinical evidence demonstrating that antigen-presenting cells educate the adaptive immune system towards an anti-inflammatory response when allergen is seen in the presence of VD3.

ELIGIBILITY:
Inclusion Criteria (study object):

1. Signed informed consent
2. Age ≥18 ≤ 60 years
3. Allergic rhinitis/rhino-conjunctivitis related to birch pollen with or without concomitant mild to moderate persistent asthma based on relative symptoms and allergy tests.
4. A positive SPT (mean wheal diameter ≥ 3mm compared to negative control and negative control should be negative) for birch pollen assessed within 1 year before randomization OR a positive serum specific anti-birch IgE-test (>0.7 U/ml)

Inclusion Criteria (healthy control):

1. Signed informed consent
2. Age, gender and location matched to a study subject. An age matched control is defined as the age of the study subject ±5 years.
3. No history of respiratory allergies and no nasal symptoms at screening.
4. A negative SPT (a positive outcome is defined as a mean wheal diameter ≥ 3mm compared to negative control and negative control should be negative) assessed within 1 year before randomization OR a negative serum specific IgE test for aeroallergens.

Exclusion Criteria:

1. A history of allergen-specific immunotherapy (SCIT or SLIT) with any allergen(s) within the 5 years before inclusion/screening visit.
2. Treatment with parenteral Vitamin D3 analogue in the year before inclusion
3. Significant, ongoing nasal symptoms caused by other allergens at study onset
4. A history of Hypercalcemia, Hypophosphatemia or vitamin D toxicity
5. Any vaccination within one week before randomization
6. Treatment with experimental products within the last 3 months or during the study or biologicals (including anti-IgE or TNF- α treatment) within the last 6 months or during the study
7. Severe immune disorders (including auto-immune diseases) and/or diseases requiring immunosuppressive drugs
8. Uncontrolled asthma or other active respiratory diseases
9. Malignancies or any malignant disease during the previous 5 years
10. Severe uncontrolled diseases that could increase the risk for subjects participating in the study, including but not limited to: cardiovascular insufficiency, any severe or unstable lung diseases, endocrine diseases, clinically significant renal or hepatic diseases, or hematological disorders
11. Active inflammation or infection of the target organs (nose, eyes or lower airways) at the start of the study
12. Use of preparations containing calcium or magnesium such as thiazide, diuretics, antacides.
13. Use of systemic steroids within 4 weeks before screening and during the study
14. Daily use of ketoconazole cream or immunosuppressive creams at planned injection site less than 7 days before or during the study
15. Pregnancy, lactation or inadequate contraceptive measures for women of child-bearing age (adequate contraceptive measures will be the use of a contraceptive device or -pill)
16. Any clinically significant abnormal laboratory parameter at screening
17. Any physical or mental condition that precludes compliance or participation in a clinical trial
18. Subjects who are employees or students of the institution or 1st grade relatives or partners of the investigators

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2015-10; Primary Completion 2016-04 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
change in IL-10 production from baseline | baseline and 4 weeks of treatment
  Compare the change in IL-10 production as marker of the induction of a more anti-inflammatory systemic immune response, at baseline and after 4 weeks of treatment comparing birch pollen allergic subjects and healthy controls in a placebo-controlled design.
change in IL-10 production from baseline | baseline and follow-up visit (between 5-7 weeks)
  Compare the change in IL-10 production as marker of the induction of a more anti-inflammatory systemic immune response, at baseline and at follow-up (between 5-7 weeks) comparing birch pollen allergic subjects and healthy controls in a placebo-controlled design.

SECONDARY OUTCOMES:
Change in IgE responses to birch pollen compared to baseline | Baseline compared to 4 weeks of treatment
  IgE responses to birch pollen measured in serum by ImmunoCAPwill be compared between subjects treated with Vitamin D3 or placebo
To evaluate the number of patients that reported adverse events with Zemplar compared to placebo. This includes adverse measurements in blood safety biochemistry/haematology parameters, urinalysis, vital signs and ECG, lung function compared to placebo. | Throughout the study and follow-up (a maximum total of 8 weeks)
  To evaluate the number of patients that reported adverse events with the VD3 analogue Zemplar® compared to placebo. This includes adverse measurements in blood safety biochemistry/haematology parameters, urinalysis, vital signs and ECG, lung function compared to placebo.
changes in percentage Th1 cells characterized by the expression of CD4, CXCR3, CCR6 and T-bet, compared to baseline | Baseline compared to 4 weeks of treatment
  Part of characterization of cellular composition with respect to T-cell subsets, B-cells and APCs
changes in percentage Th1 cells characterized by the expression of CD4, CXCR3, CCR6 and T-bet, compared to baseline | baseline and follow-up visit (between 5-7 weeks)
  Part of characterization of cellular composition with respect to T-cell subsets, B-cells and APCs
changes in percentage Th2 cells characterized by the expression of CD4, CRTh2, CCR4 and Gata-3, compared to baseline | Baseline compared to 4 weeks of treatment
  Part of characterization of cellular composition with respect to T-cell subsets, B-cells and APCs
changes in percentage Th2 cells characterized by the expression of CD4, CRTh2, CCR4 and Gata-3, compared to baseline | baseline and follow-up visit (between 5-7 weeks)
  Part of characterization of cellular composition with respect to T-cell subsets, B-cells and APCs
changes in percentage Th17/Th22 cells characterized by the expression of CD4, CCR6, CCR4, CCR10 and RORc2 compared to baseline | Baseline compared to 4 weeks of treatment
  Part of characterization of cellular composition with respect to T-cell subsets, B-cells and APCs
changes in percentage Th17/Th22 cells characterized by the expression of CD4, CCR6, CCR4, CCR10 and RORc2 compared to baseline | baseline and follow-up visit (between 5-7 weeks)
  Part of characterization of cellular composition with respect to T-cell subsets, B-cells and APCs
changes in percentage Treg cells characterized by the expression of CD4, CD25, CD127, and Foxp3 compared to baseline | Baseline compared to 4 weeks of treatment
  Part of characterization of cellular composition with respect to T-cell subsets, B-cells and APCs
changes in percentage Treg cells characterized by the expression of CD4, CD25, CD127, and Foxp3 compared to baseline | baseline and follow-up visit (between 5-7 weeks)
  Part of characterization of cellular composition with respect to T-cell subsets, B-cells and APCs
changes in percentage B cells characterized by the expression of CD19, CD5, CD20, CD27, and CD38 compared to baseline | Baseline compared to 4 weeks of treatment
  Part of characterization of cellular composition with respect to T-cell subsets, B-cells and APCs
changes in percentage B cells characterized by the expression of CD19, CD5, CD20, CD27, and CD38 compared to baseline | baseline and follow-up visit (between 5-7 weeks)
  Part of characterization of cellular composition with respect to T-cell subsets, B-cells and APCs
changes in percentage antigen presenting cells characterized by the expression of CD11c, HLA-DR, CD14, CD16, CD1c, CD141, CD123, CD19, CD163, CD68, CD86 and CD83 compared to baseline | Baseline compared to 4 weeks of treatment
  Part of characterization of cellular composition with respect to T-cell subsets, B-cells and APCs
changes in percentage antigen presenting cells characterized by the expression of CD11c, HLA-DR, CD14, CD16, CD1c, CD141, CD123, CD19, CD163, CD68, CD86 and CD83 compared to baseline | baseline and follow-up visit (between 5-7 weeks)
  Part of characterization of cellular composition with respect to T-cell subsets, B-cells and APCs
Changes in the ability of PBMCs stimulated with Bet v 1, to enhance T-cell proliferation compared to baseline | Baseline compared to 4 weeks of treatment
  PBMCs from subjects treated with Vitamin D3 or placebo will be stimulated by allergen and T-cell proliferation will be measured by looking at H3-Thymidine incorporation (measured in cpm- in counts per minute)
Changes in the ability of PBMCs stimulated with Bet v 1, to enhance T-cell proliferation compared to baseline | baseline and follow-up visit (between 5-7 weeks)
  PBMCs from subjects treated with Vitamin D3 or placebo will be stimulated by allergen and T-cell proliferation will be measured by looking at H3-Thymidine incorporation (measured in cpm- in counts per minute)
Changes in the ability of PBMCs stimulated with Bet v 1, to produce IL-5 compared to baseline | Baseline compared to 4 weeks of treatment
  PBMCs from subjects treated with Vitamin D3 or placebo will be stimulated by Bet v 1 and cytokine production will be measured (in pg/ml)
Changes in the ability of PBMCs stimulated with Bet v 1, to produce IL-5 compared to baseline | baseline and follow-up visit (between 5-7 weeks)
  PBMCs from subjects treated with Vitamin D3 or placebo will be stimulated by Bet v 1 and cytokine production will be measured (in pg/ml)
Changes in the ability of PBMCs stimulated with Bet v 1, to produce IL-13 compared to baseline | Baseline compared to 4 weeks of treatment
  PBMCs from subjects treated with Vitamin D3 or placebo will be stimulated by Bet v 1 and cytokine production will be measured (in pg/ml)
Changes in the ability of PBMCs stimulated with Bet v 1, to produce IL-13 compared to baseline | baseline and follow-up visit (between 5-7 weeks)
  PBMCs from subjects treated with Vitamin D3 or placebo will be stimulated by Bet v 1 and cytokine production will be measured (in pg/ml)
Changes in the ability of PBMCs stimulated with Bet v 1, to produce IL-17 compared to baseline | Baseline compared to 4 weeks of treatment
  PBMCs from subjects treated with Vitamin D3 or placebo will be stimulated by Bet v 1 and cytokine production will be measured (in pg/ml)
Changes in the ability of PBMCs stimulated with Bet v 1, to produce IL-17 compared to baseline | baseline and follow-up visit (between 5-7 weeks)
  PBMCs from subjects treated with Vitamin D3 or placebo will be stimulated by Bet v 1 and cytokine production will be measured (in pg/ml)
Changes in the ability of PBMCs stimulated with Bet v 1, to produce IL-10 compared to baseline | Baseline compared to 4 weeks of treatment
  PBMCs from subjects treated with Vitamin D3 or placebo will be stimulated by Bet v 1 and cytokine production will be measured (in pg/ml)
Changes in the ability of PBMCs stimulated with Bet v 1, to produce IL-10 compared to baseline | baseline and follow-up visit (between 5-7 weeks)
  PBMCs from subjects treated with Vitamin D3 or placebo will be stimulated by Bet v 1 and cytokine production will be measured (in pg/ml)
Changes in the ability of PBMCs stimulated with Bet v 1, to produce IL-21 compared to baseline | Baseline compared to 4 weeks of treatment
  PBMCs from subjects treated with Vitamin D3 or placebo will be stimulated by Bet v 1 and cytokine production will be measured (in pg/ml)
Changes in the ability of PBMCs stimulated with Bet v 1, to produce IL-21 compared to baseline | baseline and follow-up visit (between 5-7 weeks)
  PBMCs from subjects treated with Vitamin D3 or placebo will be stimulated by Bet v 1 and cytokine production will be measured (in pg/ml)
Changes in the ability of PBMCs stimulated with Bet v 1, to produce IL-22 compared to baseline | Baseline compared to 4 weeks of treatment
  PBMCs from subjects treated with Vitamin D3 or placebo will be stimulated by Bet v 1 and cytokine production will be measured (in pg/ml)
Changes in the ability of PBMCs stimulated with Bet v 1, to produce IL-22 compared to baseline | baseline and follow-up visit (between 5-7 weeks)
  PBMCs from subjects treated with Vitamin D3 or placebo will be stimulated by Bet v 1 and cytokine production will be measured (in pg/ml)
Changes in the ability of PBMCs stimulated with Bet v 1, to produce IFN-y compared to baseline | Baseline compared to 4 weeks of treatment
  PBMCs from subjects treated with Vitamin D3 or placebo will be stimulated by Bet v 1 and cytokine production will be measured (in pg/ml)
Changes in the ability of PBMCs stimulated with Bet v 1, to produce IFN-y compared to baseline | baseline and follow-up visit (between 5-7 weeks)
  PBMCs from subjects treated with Vitamin D3 or placebo will be stimulated by Bet v 1 and cytokine production will be measured (in pg/ml)
Changes in the ability of PBMCs stimulated with Bet v 1, to produce TGF-b compared to baseline | Baseline compared to 4 weeks of treatment
  PBMCs from subjects treated with Vitamin D3 or placebo will be stimulated by Bet v 1 and cytokine production will be measured (in pg/ml)
Changes in the ability of PBMCs stimulated with Bet v 1, to produce TGF-b compared to baseline | baseline and follow-up visit (between 5-7 weeks)
  PBMCs from subjects treated with Vitamin D3 or placebo will be stimulated by Bet v 1 and cytokine production will be measured (in pg/ml)
Changes in the ability of PBMCs stimulated polyclonally (anti-CD3/anti-CD28), to enhance T-cell proliferation compared to baseline | Baseline compared to 4 weeks of treatment
  PBMCs from subjects treated with Vitamin D3 or placebo will be stimulated by (anti-CD3/anti-CD28) and T-cell proliferation will be measured by looking at H3-Thymidine incorporation (measured in cpm- in counts per minute)
Changes in the ability of PBMCs stimulated polyclonally (anti-CD3/anti-CD28), to enhance T-cell proliferation compared to baseline | baseline and follow-up visit (between 5-7 weeks)
  PBMCs from subjects treated with Vitamin D3 or placebo will be stimulated by (anti-CD3/anti-CD28) and T-cell proliferation will be measured by looking at H3-Thymidine incorporation (measured in cpm- in counts per minute)
Changes in the ability of PBMCs stimulated polyclonally (anti-CD3/anti-CD28), to produce IL-5 compared to baseline | Baseline compared to 4 weeks of treatment
  PBMCs from subjects treated with Vitamin D3 or placebo will be stimulated by (anti-CD3/anti-CD28) and cytokine production will be measured (in pg/ml)
Changes in the ability of PBMCs stimulated polyclonally (anti-CD3/anti-CD28), to produce IL-5 compared to baseline | baseline and follow-up visit (between 5-7 weeks)
  PBMCs from subjects treated with Vitamin D3 or placebo will be stimulated by (anti-CD3/anti-CD28) and cytokine production will be measured (in pg/ml)
Changes in the ability of PBMCs stimulated polyclonally (anti-CD3/anti-CD28), to produce IL-13 compared to baseline | Baseline compared to 4 weeks of treatment
  PBMCs from subjects treated with Vitamin D3 or placebo will be stimulated by (anti-CD3/anti-CD28) and cytokine production will be measured (in pg/ml)
Changes in the ability of PBMCs stimulated polyclonally (anti-CD3/anti-CD28), to produce IL-13 compared to baseline | baseline and follow-up visit (between 5-7 weeks)
  PBMCs from subjects treated with Vitamin D3 or placebo will be stimulated by (anti-CD3/anti-CD28) and cytokine production will be measured (in pg/ml)
Changes in the ability of PBMCs stimulated polyclonally (anti-CD3/anti-CD28), to produce IL-17 compared to baseline | Baseline compared to 4 weeks of treatment
  PBMCs from subjects treated with Vitamin D3 or placebo will be stimulated by (anti-CD3/anti-CD28) and cytokine production will be measured (in pg/ml)
Changes in the ability of PBMCs stimulated polyclonally (anti-CD3/anti-CD28), to produce IL-17 compared to baseline | baseline and follow-up visit (between 5-7 weeks)
  PBMCs from subjects treated with Vitamin D3 or placebo will be stimulated by (anti-CD3/anti-CD28) and cytokine production will be measured (in pg/ml)
Changes in the ability of PBMCs stimulated polyclonally (anti-CD3/anti-CD28), to produce IFN-y, compared to baseline | Baseline compared to 4 weeks of treatment
  PBMCs from subjects treated with Vitamin D3 or placebo will be stimulated by (anti-CD3/anti-CD28) and cytokine production will be measured (in pg/ml)
Changes in the ability of PBMCs stimulated polyclonally (anti-CD3/anti-CD28), to produce IFN-y compared to baseline | baseline and follow-up visit (between 5-7 weeks)
  PBMCs from subjects treated with Vitamin D3 or placebo will be stimulated by (anti-CD3/anti-CD28) and cytokine production will be measured (in pg/ml)
Changes in the ability of PBMCs stimulated polyclonally (anti-CD3/anti-CD28), to produce IL-10 compared to baseline | Baseline compared to 4 weeks of treatment
  PBMCs from subjects treated with Vitamin D3 or placebo will be stimulated by (anti-CD3/anti-CD28) and cytokine production will be measured (in pg/ml)
Changes in the ability of PBMCs stimulated polyclonally (anti-CD3/anti-CD28), to produce IL-10 compared to baseline | baseline and follow-up visit (between 5-7 weeks)
  PBMCs from subjects treated with Vitamin D3 or placebo will be stimulated by (anti-CD3/anti-CD28) and cytokine production will be measured (in pg/ml)
Changes in the ability of PBMCs stimulated polyclonally (anti-CD3/anti-CD28), to produce IL-21 compared to baseline | Baseline compared to 4 weeks of treatment
  PBMCs from subjects treated with Vitamin D3 or placebo will be stimulated by (anti-CD3/anti-CD28) and cytokine production will be measured (in pg/ml)
Changes in the ability of PBMCs stimulated polyclonally (anti-CD3/anti-CD28), to produce IL-21 compared to baseline | baseline and follow-up visit (between 5-7 weeks)
  PBMCs from subjects treated with Vitamin D3 or placebo will be stimulated by (anti-CD3/anti-CD28) and cytokine production will be measured (in pg/ml)
Changes in the ability of PBMCs stimulated polyclonally (anti-CD3/anti-CD28), to produce IL-22 compared to baseline | Baseline compared to 4 weeks of treatment
  PBMCs from subjects treated with Vitamin D3 or placebo will be stimulated by (anti-CD3/anti-CD28) and cytokine production will be measured (in pg/ml)
Changes in the ability of PBMCs stimulated polyclonally (anti-CD3/anti-CD28), to produce IL-22 compared to baseline | baseline and follow-up visit (between 5-7 weeks)
  PBMCs from subjects treated with Vitamin D3 or placebo will be stimulated by (anti-CD3/anti-CD28) and cytokine production will be measured (in pg/ml)
Changes in the ability of PBMCs stimulated polyclonally (anti-CD3/anti-CD28), to produce TGF-b compared to baseline | Baseline compared to 4 weeks of treatment
  PBMCs from subjects treated with Vitamin D3 or placebo will be stimulated by (anti-CD3/anti-CD28) and cytokine production will be measured (in pg/ml)
Changes in the ability of PBMCs stimulated polyclonally (anti-CD3/anti-CD28), to produce TGF-b compared to baseline | baseline and follow-up visit (between 5-7 weeks)
  PBMCs from subjects treated with Vitamin D3 or placebo will be stimulated by (anti-CD3/anti-CD28) and cytokine production will be measured (in pg/ml)
Changes in the ability of PBMCs stimulated with PMA/Ionomycin, to produce IFN-y compared to baseline | Baseline compared to 4 weeks of treatment
  PBMCs from subjects treated with Vitamin D3 or placebo will be stimulated by PMA/Ionomycin and the percentage of cytokine producing cells will be measured as well as mean fluorescence intensity (MFI)
Changes in the ability of PBMCs stimulated with PMA/Ionomycin, to produce IFN-y compared to baseline | baseline and follow-up visit (between 5-7 weeks)
  PBMCs from subjects treated with Vitamin D3 or placebo will be stimulated by PMA/Ionomycin and the percentage of cytokine producing cells will be measured as well as mean fluorescence intensity (MFI)
Changes in the ability of PBMCs stimulated with PMA/Ionomycin, to produce IL-4 compared to baseline | Baseline compared to 4 weeks of treatment
  PBMCs from subjects treated with Vitamin D3 or placebo will be stimulated by PMA/Ionomycin and the percentage of cytokine producing cells will be measured as well as mean fluorescence intensity (MFI)
Changes in the ability of PBMCs stimulated with PMA/Ionomycin, to produce IL-4 compared to baseline | baseline and follow-up visit (between 5-7 weeks)
  PBMCs from subjects treated with Vitamin D3 or placebo will be stimulated by PMA/Ionomycin and the percentage of cytokine producing cells will be measured as well as mean fluorescence intensity (MFI)
Changes in the ability of PBMCs stimulated with PMA/Ionomycin, to produce IL-9 compared to baseline | Baseline compared to 4 weeks of treatment
  PBMCs from subjects treated with Vitamin D3 or placebo will be stimulated by PMA/Ionomycin and the percentage of cytokine producing cells will be measured as well as mean fluorescence intensity (MFI)
Changes in the ability of PBMCs stimulated with PMA/Ionomycin, to produce IL-9 compared to baseline | baseline and follow-up visit (between 5-7 weeks)
  PBMCs from subjects treated with Vitamin D3 or placebo will be stimulated by PMA/Ionomycin and the percentage of cytokine producing cells will be measured as well as mean fluorescence intensity (MFI)
Changes in the ability of PBMCs stimulated with PMA/Ionomycin, to produce IL-13 compared to baseline | Baseline compared to 4 weeks of treatment
  PBMCs from subjects treated with Vitamin D3 or placebo will be stimulated by PMA/Ionomycin and the percentage of cytokine producing cells will be measured as well as mean fluorescence intensity (MFI)
Changes in the ability of PBMCs stimulated with PMA/Ionomycin, to produce IL-13 compared to baseline | baseline and follow-up visit (between 5-7 weeks)
  PBMCs from subjects treated with Vitamin D3 or placebo will be stimulated by PMA/Ionomycin and the percentage of cytokine producing cells will be measured as well as mean fluorescence intensity (MFI)
Changes in the ability of PBMCs stimulated with PMA/Ionomycin, to produce IL-17A compared to baseline | Baseline compared to 4 weeks of treatment
  PBMCs from subjects treated with Vitamin D3 or placebo will be stimulated by PMA/Ionomycin and the percentage of cytokine producing cells will be measured as well as mean fluorescence intensity (MFI)
Changes in the ability of PBMCs stimulated with PMA/Ionomycin, to produce IL-17A compared to baseline | baseline and follow-up visit (between 5-7 weeks)
  PBMCs from subjects treated with Vitamin D3 or placebo will be stimulated by PMA/Ionomycin and the percentage of cytokine producing cells will be measured as well as mean fluorescence intensity (MFI)
Changes in the ability of PBMCs stimulated with PMA/Ionomycin, to produce IL-21 compared to baseline | Baseline compared to 4 weeks of treatment
  PBMCs from subjects treated with Vitamin D3 or placebo will be stimulated by PMA/Ionomycin and the percentage of cytokine producing cells will be measured as well as mean fluorescence intensity (MFI)
Changes in the ability of PBMCs stimulated with PMA/Ionomycin, to produce IL-21 compared to baseline | baseline and follow-up visit (between 5-7 weeks)
  PBMCs from subjects treated with Vitamin D3 or placebo will be stimulated by PMA/Ionomycin and the percentage of cytokine producing cells will be measured as well as mean fluorescence intensity (MFI)
Changes in the ability of PBMCs stimulated with PMA/Ionomycin, to produce IL-22 compared to baseline | Baseline compared to 4 weeks of treatment
  PBMCs from subjects treated with Vitamin D3 or placebo will be stimulated by PMA/Ionomycin and the percentage of cytokine producing cells will be measured as well as mean fluorescence intensity (MFI)
Changes in the ability of PBMCs stimulated with PMA/Ionomycin, to produce IL-22 compared to baseline | baseline and follow-up visit (between 5-7 weeks)
  PBMCs from subjects treated with Vitamin D3 or placebo will be stimulated by PMA/Ionomycin and the percentage of cytokine producing cells will be measured as well as mean fluorescence intensity (MFI)

CONTACTS AND LOCATIONS:
Overall Officials: Wytske J Fokkens, Prof MD PhD, Principal Investigator — Academic Medical Centre
Locations (1):
- Academic medical center, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided
The investigators have to discuss this within theEU project.